CLINICAL TRIAL: NCT00724412
Title: Evaluate Artificial Tear Efficacy in Moderate to Severe Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMA-07-15
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Dry Eye; Corneal Staining
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane (Active Comparator): Systane
  Interventions: Other: Systane
- Optive (Active Comparator): Optive
  Interventions: Other: Optive

INTERVENTIONS:
Other: Systane — Dry Eye relief eye drops
  Arms: Systane
Other: Optive — Dry Eye relief eye drops
  Arms: Optive

SUMMARY:
Comparison of two Dry Eye products

ELIGIBILITY:
Inclusion:

* Have a score of at least 2 ("some of the time") on the subject-assessed Symptom Eligibility question; see Section 8.5.1.
* Have a sodium fluorescein corneal staining sum of ≥ 3 in either eye; see Section 8.5.10.
* Have a best-corrected visual acuity of 0.6 log MAR or better in each eye as assessed using an ETDRS chart; see Section 8.5.7.

Exclusion:

* Have a history or current evidence of the following: epithelial herpes simplex keratitis (dendrictic keratitisis); vaccinia, active or recent varicella viral disease of the cornea and/or conjunctiva; ocular rosacea; acute or chronic bacterial disease of the cornea and/or conjunctiva and/or eyelids; mycobacterial infection of the eye; and/or fungal disease of the eye.
* Use of Restasis® (cyclosporine ophthalmic emulsion, 0.05%) within 30 days of Visit 1.
* Use of systemic medications that may contribute to dry eye if the dosing regimen has not been stable for at least 30 days prior to Visit
* Additionally, the dosing regimen must remain stable throughout the study period. Medications known to contribute to dry eye include, but are not limited to, cold and allergy treatments, tricyclic antidepressants, and hormone replacement therapies.
* Presence of ocular conditions such as active acute blepharitis, conjunctival infections, iritis, or any other ocular condition that may preclude the safe administration of the test article.
* Unwilling to discontinue contact lens wear at least 7 days prior to Visit 1 and during the study period.
* Current punctal occlusion of any type (e.g., collagen plugs, silicone plugs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Tear Break-up time | 42 days